CLINICAL TRIAL: NCT03439605
Title: Investigation Into the Effect of in Vitro Haemolysis on Serum High Sensitivity Troponin T Measurement, and the Determination of an Acceptable Haemolysis Index Limit
Brief Title: Effect of in Vitro Haemolysis on Serum High Sensitivity Troponin T Measurements From Patients in Accident & Emergency
Status: Completed | Type: Observational
Sponsor: Poole Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SP170327
Record Dates: First submitted 2018-02-05; First posted 2018-02-20 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Troponin T; Hemolysis
Keywords: Troponin-T; Haemolysis
MeSH Terms: conditions — Hemolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will be investigating how a common blood test for identifying heart damage (Troponin T) is affected by red blood cell damage in the blood sample (Haemolysis). It is already known that damage to the red blood cells during or after blood sample collection can cause falsely low test results however the exact amount is not clear. Some previous studies suggest that a much higher amount of red blood cell damage could be allowable when reporting the test results. This study will mimic the type of red blood cell damage that occurs in the hospital and determine what degree of damage or 'haemolysis' causes a significant reduction in the test result and therefore determine an allowable limit for safely reporting the test result. The results of this study may help provide an evidence based approach to improving current practice and may lead to fewer rejected blood samples, fewer repeat tests, improved A&E treatment times, general cost savings and an improved service to patients.

DETAILED DESCRIPTION:
This study will be investigating how a common blood test for identifying heart damage (Troponin T) is affected by red blood cell damage in the blood sample (Haemolysis). It is already known that damage to the red blood cells during or after blood sample collection can cause falsely low test results however the exact amount is not clear. Some previous studies suggest that a much higher amount of red blood cell damage could be allowable when reporting the test results. This study will mimic the type of red blood cell damage that occurs in the hospital and determine what degree of damage or 'haemolysis' causes a significant reduction in the test result and therefore determine an allowable limit for safely reporting the test result. The results of this study may help provide an evidence based approach to improving current practice and may lead to less rejected blood samples, fewer repeat tests, improved treatment times in Accident and Emergency (A&E), general cost savings and an improved service to patients.

This study will be conducted as a Masters research project in Biomedical sciences (Clinical Biochemistry) as well as providing evidence to evaluate current laboratory practice. Participants attending Poole Hospital accident and emergency who are already having blood samples taken for the heart damage blood test, high sensitivity Troponin T (hs-cTnT), are chosen for this study. As the participants are already having the hs-cTnT blood test performed it means the investigators will not be determining any new information about them from the tests and they are also the population that the results of the study will benefit.

Whilst the participants are having the routine blood samples taken for their medical investigation, an extra two blood samples will be collected (a maximum of 9 ml; less than two teaspoons) following verbal permission. Only patients with the capacity to give verbal consent will be included in the study and then their blood will only be taken once. The extra blood samples will be labelled with the time and date of collection (to ensure stability when analysing). No patient identifying information will be written on the samples and they will be sent to the laboratory in a separate bag from the routine specimens to ensure anonymity.

Once received in the laboratory, one of the study samples will be analysed for hs-cTnT and haemolysis index (a measured value that equates to the amount of haemoglobin in the sample and therefore red blood cell damage). The results from these initial tests will determine if the hs-cTnT and haemolysis are within the desired range for the study.

If the sample meets the requirements for the study, a sample specific haemolysate (Haemolysed serum) will be created from the second sample. Using both samples, varying controlled degrees of haemolysis will be created and then tested for hs-cTnT. The results from the varying degrees of haemolysis will be compared to the original unhaemolysed result to determine whether a significant change in the result has occurred.

Null hypotheses:

* There is no significant difference in hs-cTnT results between baseline and up to 100 haemolysis index. There is a significant difference in hs-cTnT results between baseline and all haemolysis index levels greater than 100.
* There is no significant difference in mean percentage change of hs-cTnT up to 100 Haemolysis index and there is a significant difference in mean percentage change of hs-cTnT at all Haemolysis levels greater than 100 haemolysis index.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients attending Poole emergency department having High Sensitivity Troponin T measurements performed on their blood as part of their medical investigations.

Exclusion Criteria:

* Serum samples with Haemolysis Index >20.
* Serum High sensitivity Troponin T result <5 ng/l and >100 ng/l
* Patients lacking capacity to give verbal consent.
* Under 18 years of age.
* Patient has previously been approached about this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients attending Poole emergency department having High Sensitivity Troponin T measurements performed on their blood as part of their medical investigations.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
The difference in measured hs-cTnT between baseline and the haemolysis groups. | Day one

SECONDARY OUTCOMES:
The Percentage change in hs-cTnT due to haemolysis at five groups of different troponin T levels. | Day one

CONTACTS AND LOCATIONS:
Locations (1):
- Poole Hospital NHSFT, Poole, Dorset, United Kingdom

IPD SHARING:
Plan to Share IPD: No